CLINICAL TRIAL: NCT03753607
Title: Changes in Doppler-derived Renal Venous Flow and Adverse Renal Outcomes Following Cardiac Surgery
Brief Title: Renal Venous Flow and Cardiac Surgery-associated Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain-Syed, Senior physician, University of Giessen
Other Study IDs: AZ 208/17 and AZ 216/17
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury; Cardiorenal Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be flash-frozen for biomarker analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The prospective single-center study investigates the association between changes in Doppler-derived renal venous flow and cardiac surgery-associated acute kidney injury (CSA-AKI).

DETAILED DESCRIPTION:
CSA-AKI is a common postoperative complication in patients undergoing open heart surgery, and is associated with increased mortality and morbidity. Venous congestion has been identified as the principal cause of cardiorenal decompensation in patients with heart failure but the relative contribution of congestion-driven renal function decline in CSA-AKI is not well studied.

The prospective single-center study investigates whether serial Doppler-derived renal venous flow assessments could help identify subset of patients with cardiorenal syndrome and subclinical renal congestion at high risk of CSA-AKI.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Subjects older than 18 years
2. Subjects undergoing elective cardiac surgery (with or without cardiopulmonary bypass)
3. Subjects who signed informed consent forms

Exclusion Criteria:

1. Patients requiring mechanical ventilation
2. Patients with mechanical circulatory assist devices or extracorporeal membrane oxygenation
3. Patients with stage 3 AKI with renal replacement therapy (RRT) or life- threatening volume overload treated with RRT
4. Stage ≥4 chronic kidney disease (CKD) stage
5. CKD requiring extracorporeal or peritoneal ultrafiltration for diuretic-resistant volume overload, 6) 6) Prediagnosed glomerulonephritis
6. Autosomal dominant polycystic kidney disease, postrenal obstruction, or solid organ transplantation
7. Anticipated life expectancy of <12 months
8. Likelihood of receiving advanced therapy (mechanical circulatory assist device/cardiac transplant)
9. Pregnancy or possibility of pregnancy in the next 3 months
10. Rhabdomyolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery (with/without cardiopulmonary bypass) at Department of Cardiovascular Surgery, University Hospital Giessen and Marburg, Campus Giessen
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Association between perioperative changes in Doppler-derived renal venous venous flow and CSA-AKI | preoperative, 24 hours postoperative, hospital discharge
  Doppler-derived renal venous flow

SECONDARY OUTCOMES:
Association of changes in postoperative renal venous flow profiles with renal recovery at hospital discharge | Measured at Day 1 and Day 7 postoperative
  Doppler-derived renal venous flow
Estimated GFR trajectory up to 3 months post-cardiac surgery relative to kidney | Measured at 3 months post-surgery
  Estimated GFR

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Böning, M.D., Study Director — University Hospital Giessen and Marburg; Horst-Walter Birk, M.D., Study Director — University Hospital Giessen and Marburg
Locations (1):
- University Hospital Giessen and Marburg-Campus Giessen, Department of Cardiovascular Surgery & Department of Nephrology, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shimada S, Hirose T, Takahashi C, Sato E, Kinugasa S, Ohsaki Y, Kisu K, Sato H, Ito S, Mori T. Pathophysiological and molecular mechanisms involved in renal congestion in a novel rat model. Sci Rep. 2018 Nov 14;8(1):16808. doi: 10.1038/s41598-018-35162-4. PMID 30429498
- [Result] Beaubien-Souligny W, Benkreira A, Robillard P, Bouabdallaoui N, Chasse M, Desjardins G, Lamarche Y, White M, Bouchard J, Denault A. Alterations in Portal Vein Flow and Intrarenal Venous Flow Are Associated With Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Cohort Study. J Am Heart Assoc. 2018 Oct 2;7(19):e009961. doi: 10.1161/JAHA.118.009961. PMID 30371304
- [Result] Iida N, Seo Y, Sai S, Machino-Ohtsuka T, Yamamoto M, Ishizu T, Kawakami Y, Aonuma K. Clinical Implications of Intrarenal Hemodynamic Evaluation by Doppler Ultrasonography in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):674-82. doi: 10.1016/j.jchf.2016.03.016. Epub 2016 May 11. PMID 27179835
- [Result] Nijst P, Martens P, Dupont M, Tang WHW, Mullens W. Intrarenal Flow Alterations During Transition From Euvolemia to Intravascular Volume Expansion in Heart Failure Patients. JACC Heart Fail. 2017 Sep;5(9):672-681. doi: 10.1016/j.jchf.2017.05.006. Epub 2017 Jul 12. PMID 28711449